CLINICAL TRIAL: NCT02210468
Title: A Phase I/II, Multicenter, Double-Blind, Placebo-controlled Safety and Efficacy Study to Evaluate APIC-CF Therapy for Mild to Moderate Primary Osteoarthritis of the Knee
Brief Title: APIC-CF Therapy for Mild to Moderate Osteoarthritis of the Knee
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cytonics Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Cyt300-01
Record Dates: First submitted 2014-07-23; First posted 2014-08-06 (Estimated); Last update posted 2015-08-21 (Estimated); Status verified 2015-08

CONDITIONS: Pain; Osteoarthritis
Keywords: Osteoarthritis; Protease Inhibitors; Alpha-2-macroglobulin; Autologous treatment; APIC-CF; Pain due to Mild to Moderate osteoarthritis (OA) of the knee
MeSH Terms: conditions — Pain; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- APIC-CF 4cc, (Experimental): APIC-CF 4cc, once at first day
  Interventions: Device: APIC-CF, 4 cc
- APIC-CF, 2cc (Experimental): APIC-CF, 2cc, one at first day
  Interventions: Device: APIC-CF, 2 cc
- Saline (Placebo Comparator)
  Interventions: Other: Placebo Comparator: Saline

INTERVENTIONS:
Device: APIC-CF, 4 cc
  Arms: APIC-CF 4cc,
Device: APIC-CF, 2 cc
  Arms: APIC-CF, 2cc
Other: Placebo Comparator: Saline — Placebo Comparator: Saline
  Arms: Saline

SUMMARY:
The mechanism of Osteoarthritis (OA) is complex, however the investigators know that cartilage breakdown follows changes in certain cells in the cartilage called chondrocytes, leading to proteases that break down cartilage. There is a protein in the human blood called alpha-2-macroglobulin that can trap these proteases and prevent the breakdown of cartilage. Cytonics developed a device that use the patient's own blood to remove all cells and concentrate alpha-2-macroglobulin to be injected in the painful knee due to osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

1. The patient provides signed written informed consent
2. The patient is willing and able to complete effectiveness and safety questionnaires and is able to read and understand study instructions in English.
3. Patient is a male or female aged between 21 - 70 years of age at the time of informed consent.
4. Patient is ambulatory (assistive devices allowed if used 4 weeks or more prior to Screening).
5. Patient has symptomatic OA in the target knee
6. Patient has a radiographic confirmation of OA at the target knee prior to screening with a grade II or III score on the K-L grading scale (Kellgren, 1957)using radiographs performed within 24 weeks of Screening
7. The patient has knee pain as demonstrated by a score of ≤3 on the KOOS pain subscale
8. The patient has venous access sufficient for APIC-CF production

Exclusion Criteria:

1. The patient has any of the following:

   * Grade 4 score on the K-L grading scale for the target knee
   * Grade 3 score on the K-L grading scale and exhibits at least one Grade 4 characteristic (large osteophytes, marked narrowing of joint space, severe sclerosis, or definite deformity of bone contour).
   * Acute fracture of the lower limb.
2. Medical history of severe bone disease (e.g., osteoporosis, osteonecrosis, joint deformity, instability, or septic arthritis).
3. The patient is categorized as grossly obese, defined as body mass index (BMI) greater than 35 kg/m2
4. Hemoglobin values <11 g/dL
5. Pregnant or breastfeeding women
6. Has clinically apparent tense effusion of the target knee.
7. Has had chondrocyte transplantation or reconstruction of ligaments in the target knee.
8. Has received an intra-articular injection(s) into any joint (e.g., corticosteroids or chondroprotective agents) within 60 days prior to Screening. Subjects receiving a corticosteroid injection during the study will be withdrawn from the study.
9. Has had surgery to the target knee within 12 months or arthroscopy of the target knee within 90 days prior to Screening.
10. Has an inflammatory disease of either knee other than OA (e.g., rheumatoid arthri septic arthritis).
11. Has another disease that can affect the health of the knee (e.g., chronic hemochromatosis; sickle cell anemia; arthropathies of systemic diseases such as chondrocalcinosis, gout, pseudogout, psoriasis, hemophilia, and infectious diseases of the joints).
12. Has significant joint infection in the target knee or inflammatory or skin disorder in the injection area of the target knee.
13. Septic arthritis in any joints within 1 year prior to screening;
14. Has fibromyalgia, anserine bursitis, lumbar radiculopathy, neurogenic or vascular claudication, vascular insufficiency of lower limbs, or peripheral neuropathy severe enough to interfere with the study evaluations.
15. Patella femoral instability
16. Patients with a history of cartilage allograft, autograft or microfracture in the study knee
17. Patients with a history of any type of blood coagulation or bleeding disorder, currently taking warfarin or other parental anticoagulant therapy or history of DVT/PE during <1 year of Screening.
18. Has a systemic or other disease or significant liver function test result from screening that, in the opinion of the investigator, would interfere with study evaluation or have an impact on the balance of benefits and risks of study treatment.
19. Diseases that may interfere:

    * type 1 diabetes
    * immunodeficiency syndrome
    * significant cardiovascular, renal, or liver disease
    * severe anemia
    * severe thrombocytopenia
    * severe infectious disease with or without fever.
    * any significant chronic skin disorders, active skin or soft tissue infection that could interfere with the evaluation of the injection site.
    * mal-alignment/deformity of the leg
    * active asthma that may require periodic treatment with steroids during the study period
    * active malignancy receiving treatment, or prior history of any malignancy, with the exception of basal cell carcinoma of the skin treated more than 1 year ago
20. Patients with psychiatric or neurological disorders including cognitive impairment or inability to provide informed consent
21. Incarcerated or confined patients
22. Medical-legal, personal injury, ongoing litigation or worker's compensation claim
23. History of drug abuse
24. Use of investigational drug, device, or biologic within 12 weeks of screening
25. Any condition that, in the opinion of the investigator, might interfere with the evaluation of the study objectives.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2015-05; Primary Completion 2016-07 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Reduction in pain after 8 weeks | 8 weeks
  Statistically significant reduction in pain after 8 weeks from initial treatment of APIC-CF compared to control as determined by the Knee injury and Osteoarthritis Outcome Score (KOOS) total score
Reduction in pain while walking at 8 weeks | 8 weeks
  Statistically significant reduction in pain while walking after 8 weeks from initial treatment of APIC-CF compared to control as determined by the Knee injury and Osteoarthritis Outcome Score (KOOS) total score

SECONDARY OUTCOMES:
Reduction in pain after 2 weeks | 2 weeks
  Statistically significant reduction in pain after 2 weeks from initial treatment of APIC-CF compared to control as determined by the Knee injury and Osteoarthritis Outcome Score (KOOS) total score.
Reduction in pain while walking at 2 weeks | 2 weeks
  Statistically significant reduction in pain while walking after 2 weeks from initial treatment of APIC-CF compared to control as determined by the Knee injury and Osteoarthritis Outcome Score (KOOS) total score
Reduction in pain at 24 weeks | 24 weeks
  Statistically significant reduction in pain after 24 weeks from initial treatment of APIC-CF compared to control as determined by the Knee injury and Osteoarthritis Outcome Score (KOOS) total score
Reduction in pain while walking after 24 weeks | 24 week
  Statistically significant reduction in pain while walking after 24 weeks from initial treatment of APIC-CF compared to control as determined by the Knee injury and Osteoarthritis Outcome Score (KOOS) total score

CONTACTS AND LOCATIONS:
Locations (1):
- IRC Clinical, Townsend, Maryland, United States